CLINICAL TRIAL: NCT04089995
Title: Coats Plus Syndrome and LCC Syndrome: Series of 10 Pediatric Cases. Review of Literature and Natural History
Acronym: COATS+
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI19_0032 (COATS+)
Record Dates: First submitted 2019-07-16; First posted 2019-09-16 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Coats Disease
Keywords: Coats; leukencephalopathy with calcifications and cysts
MeSH Terms: conditions — Retinal Telangiectasis; Cysts | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coats + and LCC syndrome
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — No intervention

SUMMARY:
Coats plus syndrome is a very rare and serious disease, caused by premature telomere shortening. It is a pediatric, multi-systemic disease, the main features of which are retinal vasculopathy and neurological disorders, associated with brain calcification and leukodystrophy. Its precise genetic etiology was discovered in 2012: autosomal recessive mutation of the CTC1 gene.

Publications about this syndrome are very few, and consist only of case reports, or small series of cases. This is explained by the rarity of occurrence of this syndrome. Since 1988, 57 cases of Coats plus syndrome have been published, with case series of up to 13 patients. Only 28 cases were detailed concerning the precise clinical presentation in the literature.

The general characteristics of this syndrome are known and, in addition to the ophthalmological and neurological damage, the various publications have been able to report a digestive attack (hemorrhages), hematological damage (central cytopenias), or increased bone fragility. No treatment is currently available to cure patients.

The natural history of this disease is poorly known. However, the most accurate knowledge possible of this disease, and its natural history, is essential. It would allow an easier identification of this rare syndrome, the establishment of a management (monitoring and therapeutic) adapted, and a more accurate genetic counseling in case of need of a prenatal diagnosis.

The description of a new series of unpublished cases, as well as a comprehensive review of the literature on Coats plus syndrome, will provide a more comprehensive and informed view of this disease.

Moreover, LCC syndrome (leukoencephalopathy with calcifications and cysts) is an autosomal recessive disorder linked to a mutation in the SNORD118 gene, which has the particularity of presenting the same neurological (neuro-radiological and clinical) characteristics, but without associating the others. ophthalmological and systemic disorders. It constitutes the differential radiological diagnosis of Coats plus syndrome. In this, the collection of medical data of French pediatric cases presenting this syndrome will allow a more detailed analysis of the differences and similarities between these two syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Coats plus genetic and / or clinical Syndrome, pediatric onset
* Patients with genetic and / or clinical LCC syndrome, pediatric onset

Exclusion Criteria:

* Refusal of the patient or his family (oral opposition)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with Coats plus genetic and / or clinical Syndrome, pediatric onset and Patients with genetic and / or clinical LCC syndrome, pediatric onset
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : seizures Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : focal clinical abnormality Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : cognitive trouble. Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with abnormal brain imaging : exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with digestive complication : bleeding Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with digestive complication :hepatic disease Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with bone complication : osteoporosis Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with ophthalmologic complication : Coats disease Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with hair or nails abnormality Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats plus syndrome and LCC syndrome about the French pediatric patients with paediatric Coats plus syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with intra uterine growth retardation or neonatal trouble : exploratory description for each patient Any disease or complication in the medical history

SECONDARY OUTCOMES:
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : seizures Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : focal clinical abnormality Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with neurological complication : cognitive trouble. Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with abnormal brain imaging : exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with digestive complication : bleeding Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with digestive complication :hepatic disease Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  percentage of patients with bone complication : osteoporosis Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with ophthalmologic complication : Coats disease Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with hair or nails abnormality Exploratory description for each patient
Precise exploration of clinical and paraclinical description of paediatric Coats + and LCC syndrome, already described in the literature about clinical cases with paediatric Coats+ syndrome, or their differential diagnosis of LCC syndrome | through study completion, an average of 1 year
  Percentage of patients with intra uterine growth retardation or neonatal trouble : exploratory description for each patient Any disease or complication in the medical history
Estimation of the natural history of the disease for morbidity and mortality from the data of the new case series and case data from the literature : | through study completion, an average of 1 year
  Average age at first symptoms Distribution of type of first symptoms Average age at diagnostic Average age at death if applicable Average age at beginning of each organ complications (ophthalmologic, neurologic, digestive, bony, or any other) Average delay of neurological deterioration Average age
Define a neuro-radiological pattern associated with Coats plus syndrome and LCC syndrome from the imaging data in the new French series | through study completion, an average of 1 year
  Blinded interpretation of MRI and CT scan Particular attention will be done about calcifications, white matter abnormalities and cysts : presence, brain localization Exploratory description of each brain abnormality found
  % of patients presenting each abnormality found and its precise description (brain localization in particular)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hopital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - CHU de Limoges, Limoges
  - Hospices civils de Lyon, Lyon
  - Fondation Adolphe de ROTHSCHILD, Paris
  - Hopital Robert Debré, Paris
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No